CLINICAL TRIAL: NCT01427270
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Active-controlled, Parallel-group, Multicenter Trial of Oxycodone/Naloxone Controlled-release Tablets (OXN) to Assess the Analgesic Efficacy (Compared to Placebo) and the Management of Opioid-induced Constipation (Compared to Oxycodone Controlled-release Tablets (OXY)) in Opioid-experienced Subjects With Uncontrolled Moderate to Severe Chronic Low Back Pain and a History of Opioid-induced Constipation Who Require Around-the-clock Opioid Therapy
Brief Title: Analgesic Efficacy and Management of Opioid-induced Constipation (OIC) for Uncontrolled Moderate - Severe Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONU3704; 2011-005060-26 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Low Back Pain
Keywords: Low back pain; Chronic pain; Opioid; Constipation; Moderate to severe chronic low back pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Constipation | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- OXN (Experimental): Oxycodone/Naloxone controlled-release tablets (OXN)
  Interventions: Drug: Oxycodone/Naloxone controlled-release
- OXY (Active Comparator): Oxycodone HCl controlled-release tablets (OXY)
  Interventions: Drug: Oxycodone HCl controlled-release
- Placebo (Placebo Comparator): Placebo tablets to match OXN or OXY
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxycodone/Naloxone controlled-release — Oxycodone/Naloxone controlled-release tablets (10/5 - 40/20 mg) taken orally every 12 hours
  Arms: OXN
Drug: Oxycodone HCl controlled-release — Oxycodone HCl controlled-release tablets (10 - 40 mg) taken orally every 12 hours
  Other Names: OxyContin
  Arms: OXY
Drug: Placebo — Placebo tablets to match OXN or OXY taken orally every 12 hours
  Arms: Placebo

SUMMARY:
The primary objective is to assess the efficacy of oxycodone/naloxone (OXN) for the management of opioid-induced constipation (OIC) compared to oxycodone controlled-release tablets (OXY) in subjects with moderate to severe low back pain and OIC who require around-the-clock opioid therapy.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female subjects ≥ 18 years of age with moderate to severe, chronic low back pain (lasting at least several hours daily) as their predominant pain condition for at least 3 months prior to screening period;
* The low back pain must be related to nonmalignant and nonneuropathic conditions and may be with or without radiation;
* Subjects must have a self-reported history of opioid induced constipation (OIC).

Exclusion Criteria include:

* Subjects with rheumatoid arthritis or other inflammatory arthritis;
* Subjects with neuropathic conditions that have been painful or required therapy within the past 3 months;
* Subjects with evidence of significant structural abnormalities of the gastrointestinal (GI) tract or other significant conditions affecting GI motility;
* Subjects with chronic constipation not related to opioid use;
* Subjects who had surgical procedures directed towards the source of chronic low back pain within 6 months of the screening visit or planned during the study;
* Subjects with a history of malignancy within the past 2 years, with the exception of basal cell carcinoma that has been successfully treated.

Other protocol specific inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall complete spontaneous bowel movement (CSBM) responder rates | Weeks 1 through 12
  The overall Complete Spontaneous Bowel Movement (CSBM) responder rates over the 12 week double-blind period comparing OXN to OXY

SECONDARY OUTCOMES:
CSBM Responder at least 50% of the weeks in the double-blind period | Weeks 1 through 12
Laxative-free Responder at least 50% of the weeks in the double-blind period | Weeks 1 through 12

CONTACTS AND LOCATIONS:
Locations (159):
- United States (140):
  - Investigational Site, Alabaster, Alabama
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Gulf Shores, Alabama
  - Investigational Site, Homewood, Alabama
  - Investigational Site, Huntsville, Alabama
  - Investigational Site, Mobile, Alabama
  - Investigational Site, Goodyear, Arizona
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Tempe, Arizona
  - Investigational Site, Tucson, Arizona
  - Investigational Site, Hot Springs, Arkansas
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Anaheim, California
  - Investigational Site, Chino, California
  - Investigational Site, Fresno, California
  - Investigational Site, Glendale, California
  - Investigational Site, La Mesa, California
  - Investigational Site, Laguna Hills, California
  - Investigational Site, Long Beach, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Los Gatos, California
  - Investigational Site, National City, California
  - Investigational Site, North Hollywood, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Paramount, California
  - Investigational Site, Richmond, California
  - Investigational Site, Roseville, California
  - Investigational Site, Sacramento, California
  - Investigational Site, San Diego, California
  - Investigational Site, Santa Ana, California
  - Investigational Site, Santa Clarita, California
  - Investigational Site, Valley Village, California
  - Investigational Site, Golden, Colorado
  - Investigational Site, New Haven, Connecticut
  - Investigational Site, Waterbury, Connecticut
  - Investigational Site, Aventura, Florida
  - Investigational Site, Boynton Beach, Florida
  - Investigational Site, Bradenton, Florida
  - Investigational Site, Clearwater, Florida
  - Investigational Site, Clermont, Florida
  - Investigational Site, Coral Gables, Florida
  - Investigational Site, Daytona Beach, Florida
  - Investigational Site, Fort Lauderdale, Florida
  - Investigational Site, Hialeah, Florida
  - Investigational Site, Inverness, Florida
  - Investigational Site, Jacksonville, Florida
  - Investigational Site, Jupiter, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Miami Lakes, Florida
  - Investigational Site, Naples, Florida
  - Investigational Site, New Port Richey, Florida
  - Investigational Site, North Miami Beach, Florida
  - Investigational Site, Orlando, Florida
  - Investigational Site, Oviedo, Florida
  - Investigational Site, Pinellas Park, Florida
  - Investigational Site, Plantation, Florida
  - Investigational Site, Port Orange, Florida
  - Investigational Site, Sanford, Florida
  - Investigational Site, South Miami, Florida
  - Investigational Site, Tamarac, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, Wellington, Florida
  - Investigational Site, Austell, Georgia
  - Investigational Site, Blue Ridge, Georgia
  - Investigational Site, Canton, Georgia
  - Investigational Site, Columbus, Georgia
  - Investigational Site, Johns Creek, Georgia
  - Investigational Site, Marietta, Georgia
  - Investigational Site, Perry, Georgia
  - Investigational Site, Savannah, Georgia
  - Investigational Site, Boise, Idaho
  - Investigational Site, Meridian, Idaho
  - Investigational Site, Bloomington, Illinois
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Evansville, Indiana
  - Investigational Site, Kansas City, Kansas
  - Investigational Site, Wichita, Kansas
  - Investigational Site, Lexington, Kentucky
  - Investigational Site, Madisonville, Kentucky
  - Investigational Site, Baton Rouge, Louisiana
  - Investigational Site, Covington, Louisiana
  - Investigational Site, Marrero, Louisiana
  - Investigational Site, Metairie, Louisiana
  - Investigational Site, Hollywood, Maryland
  - Investigational Site, Fall River, Massachusetts
  - Investigational Site, North Attleboro, Massachusetts
  - Investigational Site, Bay City, Michigan
  - Investigational Site, Pinconning, Michigan
  - Investigational Site, Rochester, Michigan
  - Investigational Site, Troy, Michigan
  - Investigational Site, Hazelwood, Missouri
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Stratford, New Jersey
  - Investigational Site, Toms River, New Jersey
  - Investigational Site, Voorhees Township, New Jersey
  - Investigational Site, Albuquerque, New Mexico
  - Investigational Site, Cedarhurst, New York
  - Investigational Site, Great Neck, New York
  - Investigational Site, New Windsor, New York
  - Investigational Site, New York, New York
  - Investigational Site, North Massapequa, New York
  - Investigational Site, Williamsville, New York
  - Investigational Site, Elkin, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Beavercreek, Ohio
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Columbus, Ohio
  - Investigational Site, Franklin, Ohio
  - Investigational Site, Groveport, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Oklahoma City, Oklahoma
  - Investigational Site, Altoona, Pennsylvania
  - Investigational Site, Jenkintown, Pennsylvania
  - Investigational Site, Johnstown, Pennsylvania
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Phoenixville, Pennsylvania
  - Investigational Site, Tipton, Pennsylvania
  - Investigational Site, Warwick, Rhode Island
  - Investigational Site, Myrtle Beach, South Carolina
  - Investigational Site, Spartanburg, South Carolina
  - Investigational Site, Franklin, Tennessee
  - Investigational Site, New Tazewell, Tennessee
  - Investigational Site, Arlington, Texas
  - Investigational Site, Athens, Texas
  - Investigational Site, Austin, Texas
  - Investigational Site, Dallas, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, Humble, Texas
  - Investigational Site, North Richland Hills, Texas
  - Investigational Site, Plano, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Sugar Land, Texas
  - Investigational Site, Tomball, Texas
  - Investigational Site, Clinton, Utah
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, West Jordan, Utah
  - Investigational Site, Richmond, Virginia
  - Investigational Site, Virginia Beach, Virginia
- Czechia (11):
  - Investigational Site, Brno
  - Investigational Site, Hradec Králové
  - Investigational Site, Most
  - Investigational Site, Olomouc
  - Investigational Site, Prague
  - Investigational Site, Praha 4 - Krc
  - Investigational Site, Rychnov nad Kněžnou
  - Investigational Site, Sternberk
  - Investigational Site, Vysoké Mýto
  - Investigational Site, Zlín
  - Investigational Site, Znojmo
- Investigational Site, Catania, Italy
- Poland (7):
  - Investigational Site, Bielsko-Biala
  - Investigational Site, Bydgoszcz
  - Investigational Site, Gdansk
  - Investigational Site, Gdynia
  - Investigational Site, Katowice
  - Investigational Site, Lublin
  - Investigational Site, Torun